CLINICAL TRIAL: NCT07031037
Title: Exploratory Study of Sensory Profile and Coping Strategies in Eating Disorders
Acronym: SensoryCop
Status: Not yet recruiting | Type: Observational
Sponsor: Centre Hospitalier Esquirol (Other)
Responsible Party: Principal Investigator, Aude Paquet, Psychomotor Therapist, Doctor in Psychology, Centre Hospitalier Esquirol
Other Study IDs: 2024-A01154-43
Record Dates: First submitted 2025-05-14; First posted 2025-06-22 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-05

CONDITIONS: Eating Disorders; Anorexia Nervosa; Boulimia Nervosa; Hyperphagia
Keywords: Sensory Profile; Coping Strategies; Eating Disorders; sensory processing disorder
MeSH Terms: conditions — Feeding and Eating Disorders; Anorexia Nervosa; Hyperphagia | interventions — Weights and Measures

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Scales — Five questionnaires were administered at inclusion, socio-demographic and clinical data were collected during an interview (anxiety-depression, treatments).
  The following questionnaires were used: The Revised Ritvo Autism and Asperger Diagnostic Scale (RAADS-R-Fr), the Eating Disorder Examination Self-Report Questionnaire (EDE-Q), the Adolescent/Adult Sensory Profile (AASP), the Coping Inventory for Stressful Situations (CISS), the Hospital anxiety and depression scale (HAD) and the Multidimensional Assessment of Interoceptive Awareness Version 2 (MAIA-2).

SUMMARY:
This descriptive study aims primarily to characterize the sensory profile of patients with eating disorders (divided into three diagnostic groups: anorexia nervosa, boulimia nervosa and hyperphagia), controlling for possible autistic traits in this population.

The study involves measuring characteristics associated with eating disorders (diagnosis, BMI, anxiety), assessing the sensory profile (AASP), and coping strategies in patients with eating disorders who are hospitalised or followed up in consultation.

ELIGIBILITY:
Inclusion Criteria:

* Gender and Age: Male or female, aged 18 to 65
* Confirmed diagnosis of anorexia nervosa (F50.01; F50.02), boulimia nervosa (F50.2), hyperphagic episodes (F50.8) or restriction or avoidance of food intake (F50.8) according to DSM-5 criteria
* Hospitalization or consultation for Eating Disorder at Centre Hospitalier Esquirol
* Consent: Free, informed, and written consent, signed by the participant and/or their legal representative (for participants under protection measures) and the investigator (at the latest on the day of inclusion and before any research-related examination).

Exclusion Criteria:

* Psychiatric comorbidity (non-tobacco addiction, characterized depressive episode, bipolar disorder, obsessive-compulsive disorder, schizophrenia and related disorders, neurodevelopmental disorder)
* History of Eating Disorder other than current disorder
* Proven sensory or neurological disability
* Inability to understand questionnaires and information related to the study
* Persons under psychiatric care in accordance with articles L. 3212-1 and L. 3213-1
* Pregnant, nursing or parturient women
* Adults subject to legal protection or unable to express their consent to express their consent
* Persons not affiliated to a social security scheme or not benefiting from one social security scheme
* Persons deprived of their liberty by judicial or administrative decision

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be enrolled during hospitalization or consultation of their Eating Disorder treatment in the Esquirol Hospital Center of Limoges, France.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2028-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Sensory profile from the Adolescent and Adult Sensory Profile (Brown and Dunn, 2002) according to each diagnostic group. | At enrollment
  Sensory profile scores will be obtained using the Adolescent and Adult Sensory Profile (AASP) scale during an individual interview after the participant has been included in the study. Subscores for sensory sensitivity, low registration, sensation seeking, and sensation avoidance will be collected. For each subscore, the minimum and maximum values range from 15 to 75. A high score indicates high sensory sensitivity.
Scores for task coping drawn from the Coping Inventory for Stressful Situations (Endler & Parker, adapted by JP Rolland) according to each diagnostic group | at enrollment
  Coping scores will be obtained using the Coping Inventory for Stressful Situations (CISS) scale during an individual interview after the participant has been included in the study. The task-oriented coping subscore, emotion subscore, avoidance subscore, distraction subscore, and social diversion subscore will be collected. The minimum and maximum values range from 16 to 90. A high score indicates high oriented coping.

SECONDARY OUTCOMES:
Description of the frequency of autistic traits for each diagnostic group | At enrollment
  The frequency of autistic traits will be obtained using the Revised Ritvo Autism and Asperger Diagnostic Scale (RAADS-R-Fr) during an individual interview after the participant has been included in the study. The minimum and maximum values range from 0 to 240. The generally accepted threshold for significant autistic traits is 70. A high score indicate high autistic traits.
Description of the frequency of eating disorders for each diagnostic group. | At enrollment
  Eating disorders will be assessed using the Eating Disorder Examination Self-Report Questionnaire (EDE-Q) during an individual interview after the participant's inclusion. The EDE-Q, provide subscale scores reflecting the severity of aspects of the psychopathology of eating disorders. The subscales are Restraint, Eating Concern, Shape Concern and Weight Concern. For Restaint subscale minimum and maximum values range from 0 to 30. For Eating Concern subscale minimum and maximum values range from 0 to 30. For Shape Concern subscale minimum and maximum values range from 0 to 48. For Weight Concern subscale minimum and maximum values range from 0 to 30.
  The higher the score, the more severe the symptoms.
Anxiety according to each diagnostic group. | At enrollment
  Anxiety and depression will be obtained using the Hospital Anxiety and Depression Scale (HAD) during an individual interview after the participant's inclusion. The anxiety subscore will be collected. Minimum and maximum values range from 0 to 21. The generally accepted threshold for significant anxiety is 11.
Body awareness from the multidimensional assessment of interoceptive awareness for each diagnostic group. | At enrollment
  Body awareness will be obtained using the Multidimensional Assessment of Interoceptive Awareness Version 2 (MAIA-2) scale during an individual interview after the participant's inclusion. Minimum and maximum values range from 0 to 185. A high score indicates high interoceptive awareness.

CONTACTS AND LOCATIONS:
Locations (1):
- Esquirol Hospital Center, Limoges, Nouvelle-Aquitaine, France

IPD SHARING:
Plan to Share IPD: No